CLINICAL TRIAL: NCT05245643
Title: STIMulation cérébrale Profonde Chez Des Patients Souffrant d'Anorexie Mentale Résistante et Sévère
Brief Title: Deep Brain Stimulation for Severe Anorexia Nervosa
Acronym: STIMARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D21-P014
Record Dates: First submitted 2021-05-26; First posted 2022-02-18 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Anorexia Nervosa
Keywords: Disease Resistance; Deep brain stimulation; Neuropsychological Tests; Patient Acceptance of Health Care
MeSH Terms: conditions — Anorexia Nervosa; Disease Resistance; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Prospective multicenter study: interventional cohort for surgical treatment (deep brain stimulation) in severe and resistant Anorexia Nervosa
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with severe and resistant Anorexia Nervosa (Other): 12 consecutive patients fulfilling the inclusion criteria and consenting to participate in the research, recruted in the three inclusion centers.
  Interventions: Device: Abbott Infinity Deep Brain Stimulation System

INTERVENTIONS:
Device: Abbott Infinity Deep Brain Stimulation System — DBS is robot-assisted, with 3D intraoperative imaging control, under general anesthesia. Target is defined thanks to preoperative dedicated MRI with 2 independent experts' assessment.
  Other Names: DBS of both nucleus accumbens

SUMMARY:
The somatic complications as well as the suicidal risk make Anorexia Nervosa (AN) the psychiatric disease with the highest mortality rate: the standardized mortality ratio is higher than 4 and 1 in 5 patients with AN who dies has committed suicide. Approximately 20% of patients suffering from AN evolves into a chronic form without prolonged remission. These patients are at high risk of serious complications (somatic and psychiatric). The peak incidence of AN lies between 15 and 19 years: patients suffering from severe and resistant AN are therefore mostly young people. At present, there is no treatment for severe and resistant AN. New insights in AN pathophysiology revealed that AN patients develop a kind of "addiction" to thinness which contributes to weight loss despite negative consequences. In parallel, Deep Brain Simulation (DBS) is now widely performed for movements disorders with good results and low morbidity. DBS is also currently under investigations for other indications such as obsessional compulsive disorder or pharmacoresistant epilepsy. Some case series reported promising results of DBS for severe and resistant AN. The aim of this study is to investigate the safety of nucleus accumbens chronic stimulation for patients enduring severe and resistant AN. Secondary objective is to evaluate patient's acceptance of this new treatment.

DETAILED DESCRIPTION:
Main objective:

To selectively target for neuromodulation the key structures known to be involved in the motivational aspect of food intake, i.e. the nucleus accumbens, while evaluating safety and tolerance in the specific setting of AN patients (monitoring of serious adverse events [SAE])

Secondary objectives:

1. Evaluation of patient's acceptance,
2. Effect of DBS on weight stabilization (maintenance of patients' BMI above 14kg/m2),
3. Effect of DBS on pupillometry in patients with severe and resistant AN,
4. Effect of DBS on intermediate clinical variables such as loss of cognitive flexibility, overestimation of delayed rewards, and central coherence defect,
5. Effect of DBS on psychiatric comorbidities of patients suffering from severe and resistant AN.

Prospective multicenter study: interventional cohort

Practical conduct:

A. If all the inclusion criteria are met, proposal to participate in the study allowing a time window of 2 weeks of reflection before giving consent, B. Joint neurosurgeon/psychiatrist information consultation with delivery of a consent form, C. Preoperative assessment carried out after a delay of at least 2 weeks (anaesthesia consultation, brain MRI and neurocognitive assessment), D. Admisison in neurosurgery for one week to perform the DBS procedure. Post-operative CT Scan. The stimulation is turned on for all patients upon discharge from the hospital , E. Joint follow-up visit with the referring physician (once a month) and the neurosurgeon (once every 2 months) for 12 months F. Two neurocognitive assessments during follow-up visit : one early and one late postoperative (respectively at 5 and 11 months)

Inclusion period: 24 months Duration of preoperative assessment and reflection phase: 3 months Duration of participation (treatment + follow-up): 12 months Total duration: 40 months

Statistical analyses:

Descriptive results are presented as means ± standard deviations for continuous data and as percentages for categorical data.

The unpaired and paired t-test because of repeated measures in the same subjects, the Fisher's exact test will be use. A p<0.05 will be considered as statistically significant. A binomial sequence test is performed after each patient inclusion to check that the rate of SAE remains inferior to 25%.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Anorexia nervosa according to DSM V criteria.
2. Age 18 to 65 years.
3. Chronic, treatment-resistant anorexia nervosa, defined as:

   * Anorexia nervosa evolving for at least 7 years.
   * Inability to maintain a BMI ≥ 17kg/m² for 2 months following hospitalization in a center specialized for the management of patients suffering from eating disorders according to the criteria of the French Federation of Anorexia and Bulimia nervosa and the Directorate General of Care Provision (Direction Générale de l'Offre de Soins - DGOS, in French). Failure of at least 2 hospitalizations in a specialized center during the history of the disease.
   * Inability to maintain a BMI ≥ 17kg/m² for more than 3 consecutive months during an outpatient treatment conducted by a team specialized for the care of patients suffering from eating disorders according to the criteria of the French Federation of Anorexia and Bulimia and the Directorate General of Care Provision (Direction Générale de l'Offre de Soins - DGOS, in French) in the year preceding the inclusion. Failure of at least 2 outpatient treatments conducted by a specialized team during the AN care.
4. Impaired psychological, social and occupational functioning defined by a score ≤ 45 on the Global Assessment of Functioning Scale.
5. Anorexia nervosa is judged to be the primary disorder if there are psychiatric comorbidities such as depression, anxiety disorder, obsessive-compulsive disorder, or personality disorder by at least two independent experts.
6. The patient is able to comply with the operational and administrative requirements of the study and is able to complete the protocol forms.
7. Patient provides written informed consent.
8. Patient is drug-free or on a medication that has been stable for at least 6 weeks at the time of study entry.
9. If female subject and of childbearing age: use of an effective method of contraception.
10. Membership in a health insurance plan or beneficiary.

Exclusion Criteria:

1. Presence of an Axis I disorder that is primary to anorexia nervosa.
2. Presence of a personality disorder that could compromise compliance with post-surgical follow-up assessed by 2 independent experts
3. Presence of severe neurological pathology or significant MRI abnormalities (excluding anorexia-related atrophy).
4. Cognitive and intellectual ability to understand the risks and constraints of the technique or to give informed consent.
5. Albumin levels <30g/L.
6. Presence of medical contraindications to undergo implantation of a DBS system or to realize an MRI (pacemaker).
7. Pregnant or breastfeeding woman.
8. Previous DBS.
9. Trusted person and/or family object to patient's participation.
10. Contraindication to general anesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Rate of serious adverse event | Through study completion (2 years)
  A serious adverse event is defined as any untoward medical occurrence that at any dose:
  Results in death Is life-threatening Requires inpatient hospitalization or causes prolongation of existing hospitalization Results in persistent or significant disability/incapacity May have caused a congenital anomaly/birth defect Requires intervention to prevent permanent impairment or damage. In this study, SAE are permanently monitored. After each patient inclusion, SAE rate is calculated: it has to remain inferior to 25% of the included population.

SECONDARY OUTCOMES:
Measure of protocol acceptability | At the end of the inclusions (2 years after study start)
  Number of patients meeting inclusion criteria and accepting treatment / Number of patients meeting inclusion criteria and offered treatment
BMI Monitoring | Through study completion (each month), during 2 years
  Variation of BMI.
Pupillometry variation | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Pupillometry according to GHU PARIS Sainte Anne Clinique des Maladies Mentales et de l'Encéphale protocol.
Scores of Eating Disorder Inventory-2 | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  The EDI consists of 8 subscales measuring drive for thinness, bulimia, body dissatisfaction, ineffectiveness, perfectionism, interpersonal distrust, interoceptive awareness, and maturity fears.
Scores of Delayed Discounting Task | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure of temporal discounting, the tendency for people to prefer smaller, immediate monetary rewards over larger, delayed rewards
Scores of The Brixton Spatial Anticipation Test | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Measures the ability to detect rules in sequences of stimuli.
Scores of the Trail Making Test | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  assess executive function
Scores of the slips-of-action task | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure habit tendencies, the likelihood of making erroneous responses for devalued outcome
Scores of the Wisconsin Card Sorting Test | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure the ability to display flexibility in the face of changing schedules of reinforcement
Scores of the Montreal Cognitive Assessment | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  screening assessment for detecting cognitive impairment
Scores of the Dubois' five words testing | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Assess the verbal episodic memory
Scores of the Rey-Osterrieth Complex Figure Test (ROCFT) | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure of constructional praxis and visual recall
Scores of the Hospital Anxiety and Depression scale | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  detect states of depression and anxiety
Scores of the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Rate the severity of obsessive-compulsive disorder symptoms
Scores of the Scale for Suicide Ideation | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Measures the current intensity of patients' specific attitudes, behaviors, and plans to commit suicide on the day of the interview.
Scores of the Short Form (36) Health Survey | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure of health status
Scores of the Global Assessment of Functioning | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Rate subjectively the social, occupational, and psychological functioning of an individual
Scores of the Zarit Burden Interview | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  Assess caregiving burden in clinical and research settings
The Taylor Complex Figure Test (TCFT) | Through study completion: during the preoperative (2 weeks before the surgery), early postoperative (1 month after the surgery), late postoperative (4 months after the surgery) and end of study (11 months after the surgery) neurocognitive assessments
  measure of constructional praxis and visual recall

CONTACTS AND LOCATIONS:
Locations (1):
- Viviane AWASSI, Paris, France

IPD SHARING:
Plan to Share IPD: No